CLINICAL TRIAL: NCT00002134
Title: A Randomized, Controlled Study of the Safety and Preventive Efficacy of Oral Ganciclovir When Used in Conjunction With An Intravitreal Ganciclovir Implant in the Treatment of Cytomegalovirus Retinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roche Global Development (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 037B; GANS2304
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-07

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; Ganciclovir; Administration, Oral; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Acquired Immunodeficiency Syndrome | interventions — Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir

SUMMARY:
To demonstrate the efficacy of oral ganciclovir in preventing new cytomegalovirus (CMV) disease in AIDS patients with unilateral CMV retinitis treated with an intravitreal ganciclovir implant. To compare safety and tolerance, time to progression, quality of life, and survival among patients treated with an intravitreal ganciclovir implant, with and without oral ganciclovir, versus standard intravenous (IV) ganciclovir therapy.

DETAILED DESCRIPTION:
Patients receive intravitreal ganciclovir implant plus oral ganciclovir, intravitreal implant alone, or IV ganciclovir.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Topical drugs and ophthalmics.

Patients must have:

* AIDS.
* Unilateral CMV retinitis.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Chronic, clinically significant diarrhea, nausea, abdominal pain,or other symptoms of uncontrolled gastrointestinal disease.
* Ocular opacities (corneal, aqueous, lens, or vitreous) preventing ophthalmologic retinal assessment of fundus photography.
* Acute retinal necrosis or any other intraocular condition that might preclude study completion.
* Ocular condition requiring immediate surgery.
* Unable to have long-term IV catheter placement.

Concurrent Medication:

Excluded:

* Vidarabine.
* Amantadine hydrochloride.
* Cytarabine.
* FIAC or FIAU.
* Idoxuridine.
* Ribavirin.
* Valacyclovir.
* Foscarnet.
* CMV hyperimmune globulin.
* Soluble CD4.
* Trichosanthin.
* Imipenem-cilastatin.
* Isoprinosine.
* Levamisole.
* Interferon.
* Other investigational drugs.

Patients with the following prior conditions are excluded:

* History of previous invasive intraocular surgery of any kind in the involved eye or any condition for which ocular surgery is contraindicated.
* History of hypersensitivity to acyclovir or ganciclovir.

Prior Medication:

Excluded:

* Any prior oral ganciclovir in a CMV retinitis treatment protocol OR more than 4 months of prior oral ganciclovir in a prophylaxis study (per amendment).
* Prior intravitreal ganciclovir implant.
* More than two prior induction dose courses of IV anti-CMV therapy (per amendment).
* Intravitreal injection of any antiviral medication within the past 4 weeks (per amendment).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Dr Neil Brourman, Beverly Hills, California
  - UCI College of Medicine, Irvine, California
  - Estelle Doheny Eye Clinic, Los Angeles, California
  - Dr Robert T Wendel, Sacramento, California
  - Kaiser Hosp, San Francisco, California
  - Pacific Horizons Med Group, San Francisco, California
  - Santa Clara Valley Med Ctr, San Jose, California
  - Dr Robert Avery, Santa Barbara, California
  - Harbor - UCLA Med Ctr, Torrance, California
  - Dr Alan Palestine, Washington D.C., District of Columbia
  - Dr Michael Stewart, Jacksonville, Florida
  - Bascom Palmer, Miami, Florida
  - Emory Eye Clinic, Atlanta, Georgia
  - Dr David Weinberg, Chicago, Illinois
  - Univ of Kentucky Med Ctr, Lexington, Kentucky
  - New England Med Ctr / Tufts Univ, Boston, Massachusetts
  - Dr Dorothy Friedberg, New York, New York
  - Saint Clare's Prof Office, New York, New York
  - New York Hosp, New York, New York
  - Vitreo - Retinal Consultants, New York, New York
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Univ of Washington Med Ctr, Seattle, Washington

REFERENCES:
- [Background] Cheng B. Guide to CMV management. PI Perspect. 1996 Apr;(no 18):13-4. PMID 11363508